CLINICAL TRIAL: NCT05644418
Title: Electrical Impedance Tomography During Flow Controlled Ventilation in the Intensive Care Unit
Brief Title: EIT During FCV in the Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Ventinova (Unknown)
Responsible Party: Principal Investigator, Henrik Endeman, H. Endeman, MD, PhD, Principle Investigator, Erasmus Medical Center
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: NL 68962.078.19
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Post-cardiac Surgery
Keywords: FCV; EIT; Mechanical Power; Minute volume; Dissipated energy; ICU

STUDY DESIGN:
Intervention Model Description: PCV at baseline, followed by 90 minutes of FCV and finished with 30 minutes of PCV
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Postcardiac surgery ICU-patients (Experimental): After postcardiac surgery patients are brought to the ICU and are ventilated on PCV (Pressure Controlled Ventilation). Measurements of the lung volume (by Electrical Impedance Tomography; EIT), the minute volume and Mechanical Power/Dissipated energy are started and continued for the duration of the study. After a few minutes the patient is switched to FCV (Flow Controlled Ventilation) for 90 minutes and afterwards PCV is resumed with the measurements lasting for another 30 minutes (total study time 120 minutes).
  Interventions: Device: Flow Controlled Ventilation (FCV)

INTERVENTIONS:
Device: Flow Controlled Ventilation (FCV) — FCV is started with the same settings as PCV (PEEP, Ppeak, FiO2) and after 30 minutes FCV is optimized concerning the driving pressure and PEEP using the dynamic compliance. After a total of 60 minutes the flow is adjusted based on the arterial blood gas.

SUMMARY:
The goal of this clinical trial is to study the effects of Flow Controlled Ventilation (FCV) following conventional mechanical ventilation (Pressure or Volume Controlled Ventilation) in postcardiac surgery ICU-patients to allow for future power calculations and to obtain experience with FCV.

The main questions it aims to answer are:

* What is the effect of FCV on the lung volume measured by Electrical Impedance Tomography (EIT)?
* What is the effect of FCV on the minute volume?
* What is the effect of FCV on the mechanical power and dissipated energy?

Participants will be ventilated with PCV at baseline and then switched to FCV for 90 minutes while the lung volume, minute volume and mechanical power and dissipated energy levels are measured.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older;
* Informed consent form signed by the subject or a legal representative;
* Controlled mechanical ventilation via an endotracheal tube -
* FiO2 ≤50% and PEEP 10 cmH2O or lower

Exclusion Criteria:

* Severe sputum stasis or production requiring frequent bronchial suctioning (more than 5 times per nurse shift)
* Severe respiratory insufficiency defined as a PaO2 to FiO2 ratio of <100mmHg or moderate to severe ARDS according to the Berlin definition of ARDS
* Untreated pneumothorax (i.e. no pleural drainage)
* Hemodynamic instability defined as a mean arterial pressure below 60mmHg not responding to fluids and/or vasopressors or a noradrenalin dose >0.4mg/kg/min
* Excessive subcutaneous emphysema (prevents proper functioning of the EIT device)
* Thoracic wounds, bandages or other obstruction which prevent proper functioning of the EIT device
* High (>15 mmHg) or instable (an increase in sedation or osmotherapy is required) intracranial pressure
* An inner tube diameter of 6mm or less

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
End-expiratory lung volume | Baseline EELV compared to after 30 minutes of FCV (same ventilator settings)
  The difference in End-expiratory lung volume (EELV) between PCV and FCV is measured using the difference in End-expiratory lung impedance (EELI) and tidal volume at baseline

SECONDARY OUTCOMES:
Minute volume | The difference in minute volume between PCV at baseline and after 90 minutes of FCV (after optimization of FCV)
  The difference in minute volume between PCV and FCV with a stable PaCO2
Mechanical Power | The difference in Mechanical Power between PCV at baseline and after 90 minutes of FCV (after FCV optimization)
  The difference in Mechanical Power between PCV and FCV are measured by using our own produced Pressure-Volume loops
Dissipated energy | The difference in Dissipated energy between PCV at baseline and after 90 minutes of FCV (after FCV optimization)
  The difference in Dissipated energy between PCV and FCV are measured by using our own produced Pressure-Volume loops

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Endeman, MD, PhD, Principal Investigator — Erasmus MC, Rotterdam
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Van Oosten JP, Francovich JE, Somhorst P, van der Zee P, Endeman H, Gommers DAMPJ, Jonkman AH. Flow-controlled ventilation decreases mechanical power in postoperative ICU patients. Intensive Care Med Exp. 2024 Mar 19;12(1):30. doi: 10.1186/s40635-024-00616-9. PMID 38502268